CLINICAL TRIAL: NCT02633800
Title: Randomized, Placebo-controlled, Double-blind Phase 2 Study of Patritumab (U3-1287) in Combination With Cetuximab Plus Platinum-based Therapy in First Line Setting in Subjects With Recurrent or Metastatic Squamous Cell Carcinoma of the Head and Neck
Brief Title: Patritumab With Cetuximab and a Platinum Agent for Squamous Cell Carcinoma (Cancer) of the Head and Neck (SCCHN )
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Trial was terminated by sponsor due to lack of efficacy.
Sponsor: Daiichi Sankyo (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: U31287-A-U203; 2015-002222-40 (EudraCT Number)
Record Dates: First submitted 2015-12-15; First posted 2015-12-17 (Estimated); Results first posted 2019-01-07 (Actual); Last update posted 2019-01-07 (Actual); Status verified 2018-12

CONDITIONS: Head and Neck Neoplasms
Keywords: Squamous cell cancer of the head and neck; Squamous cell carcinoma; Head and neck cancer; Neoplasms by site
MeSH Terms: conditions — Head and Neck Neoplasms; Carcinoma, Squamous Cell; Neoplasms by Site | interventions — patritumab; Cetuximab; Cisplatin; Carboplatin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Patritumab (Experimental): All participants receive patritumab with cetuximab plus platinum-based therapy (cisplatin or carboplatin)
  Interventions: Drug: Patritumab; Drug: Cetuximab; Drug: Cisplatin; Drug: Carboplatin
- Placebo (Placebo Comparator): All participants receive placebo with cetuximab plus platinum-based therapy (cisplatin or carboplatin)
  Interventions: Drug: Cetuximab; Drug: Cisplatin; Drug: Carboplatin; Drug: Placebo

INTERVENTIONS:
Drug: Patritumab — Patritumab initial loading dose is 18 mg/kg IV over 60 minutes followed by a maintenance dose of 9 mg/kg IV over 60 minutes (± 10 minutes) every three weeks
  Other Names: U3-1287
  Arms: Patritumab
Drug: Cetuximab — Cetuximab 400 mg/mg/m^2 IV loading dose, followed by 250 mg/m^2 weekly
Drug: Cisplatin — Cisplatin at 100 mg/m^2 IV infused over 1 hour, every three weeks up to a maximum of 6 cycles
  Other Names: Platinum-based therapy
Drug: Carboplatin — Carboplatin IV over 30 to 60 minutes, every 3 weeks for a maximum of 6 cycles
  Other Names: Platinum-based therapy
Drug: Placebo — Placebo to match patritumab
  Arms: Placebo

SUMMARY:
This study will test an investigational study drug called patritumab. It is a 'randomized study' which means participants have an equal chance of being assigned to receive the experimental medication (patritumab) or a substance that looks like the experimental product, but is not (placebo). Patritumab may work when combined with other medications that are approved for the treatment of head and neck cancer. They are called cetuximab, cisplatin or carboplatin. All participants will receive the other medications approved for treatment of head and neck cancer, even if they do not receive the experimental product.

DETAILED DESCRIPTION:
Main objective of the trial:

The main objective of the trial is to evaluate progression-free survival (PFS) in the heregulin (HRG) high expression population from subjects treated with patritumab + cetuximab + platinum-based therapy compared to placebo + cetuximab + platinum-based therapy.

ELIGIBILITY:
Inclusion Criteria:

* Has histologically confirmed recurrent disease or metastatic SCCHN tumor and/or from its lymph nodal metastases originating from the oral cavity, oropharynx, hypopharynx, and larynx
* Has or be willing to provide tumor tissue for testing
* Has measurable disease per Response Evaluation Criteria in Solid Tumor (RECIST) version 1.1
* Has Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1
* Has adequate hematological function per protocol
* Has adequate renal function per protocol
* Has adequate hepatic function per protocol
* Agrees to use effective contraception while on the study and for 6-months after the end of the study
* Provides written informed consent(s)

Exclusion Criteria:

* Has left ventricular ejection fraction (LVEF) <50%
* Had prior epidermal growth factor receptor (EGFR) targeted regimen
* Had prior anti-human epidermal growth factor receptor 3 (anti-HER3) therapy
* Had prior chemotherapy for recurrent/metastatic disease
* Had anti-cancer therapy between biopsy and submission of sample
* Has history of other malignancies, except adequately treated non-melanoma skin cancer, curatively treated in-situ disease, or other solid tumors curatively treated with no evidence of disease for ≥ 2 years
* Has known history of brain metastases or active brain metastases
* Has uncontrolled hypertension
* Has clinically significant electrocardiograph (ECG) findings
* Had myocardial infarction within 1 year before enrollment, symptomatic congestive heart failure, unstable angina, or arrhythmia requiring medication
* Had platinum-containing drug therapy with radiotherapy less than 6 months before study drug treatment
* Had therapeutic or palliative radiation therapy or major surgery within 4 weeks before study drug treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 87 (Actual)
Dates: Start 2015-12-22 (Actual); Primary Completion 2018-01-11 (Actual); Study Completion 2018-02-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kevin Harrington, Prof, MD, Principal Investigator — Royal Marsden NHS Foundation Trust
Locations (34):
- Belgium (3):
  - Institut Jules Bordet, Brussels
  - Univeristair Ziekenhuis Antwerpen, Edegem
  - UZ Leuven, Leuven
- France (10):
  - Institut Curie, Paris, Cedex
  - Institut de Cancerologie de l'Ouest, Angers
  - Centre Hospitalier de Bordeaux - Hôpital Saint André, Bordeaux
  - Hopital Croix-Rousse, Lyon
  - Centre Leon Berard, Lyon
  - CHU Hopital de la Timone, Marseille
  - Hopital Saint Joseph, Marseille
  - Centre de Cancerologie du Grand Montpellier, Montpellier
  - Institut de Cancerologie de l'Ouest, Saint-Herblain
  - Gustave Roussy, Villejuif
- Germany (3):
  - Charite Universitatsmedizin Berlin, Berlin
  - Medizinische Hochschule Hannover, Hanover
  - Klinikum der Universitat Munchen, München
- Hungary (5):
  - Orszagos Onkologiai Intezet, Budapest
  - Debreceni Egyetem Orvos-es Egeszsegtudomanyi Centrum, Debrecen
  - Bacs-Kiskun Megyei Korhaz, Kecskemét
  - Borsod Abauj Zemplen Megyei Korhaz es Egyetemi Oktato Korhaz, Miskolc
  - Josa Andras Oktatokorhaz, Nyíregyháza
- Poland (3):
  - Centrum Onkologii im. Prof. Franciszka Lukaszczyka w Bydgoszczy, Bydgoszcz
  - Przychodnia Lekarska "KOMED", Konin
  - Regionalny Osrodek Onkologiczny Szpital im. M. Kopernika w Lodzi, Lodz
- Romania (3):
  - Medisprof SRL, Cluj-Napoca
  - Centrul de Oncologie Sfantul Nectarie, Craiova
  - Institutul Regional de Oncologie Iasi, Iași
- United Kingdom (7):
  - University College London Hospitals NHS Foundation Trust - University College Hospital, London
  - Guy's and St Thomas' NHS Foundation Trust - St Thomas' Hospital, London
  - The Royal Marsden NHS Foundation Trust, London
  - Weston Park Hospital, Sheffield
  - The Shrewsbury and Telford Hospital NHS Trust, Shrewsbury
  - Southampton General Hospital, Southampton
  - The Royal Marsden NHS Foundation Trust, Sutton

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) and applicable supporting clinical trial documents may be available upon request at http://www.clinicalstudydatarequest.com. In cases where clinical trial data and supporting documents are provided pursuant to our company policies and procedures, Daiichi Sankyo will continue to protect the privacy of our clinical trial participants. Details on data sharing criteria and the procedure for requesting access can be found at this web address: https://www.clinicalstudydatarequest.com/Study-Sponsors-DS-Details.aspx
Supporting Information: Study Protocol, SAP, CSR, Analytic Code
Time Frame: Studies for which the medicine and indication have received EU and US marketing approval on or after 01 January 2014 or by the US or EU Health Authorities when regulatory submissions in both regions are not planned and after the primary study results have been accepted for publication.
Access Criteria: Formal request from qualified scientific and medical researchers on IPD and clinical study documents from clinical trials supporting products submitted and licensed in the United States and the European Union from 01 January 2014 and beyond for the purpose of conducting legitimate research. This must be consistent with the principle of safeguarding study participants' privacy and consistent with provision of informed consent.
URL: https://www.clinicalstudydatarequest.com/Study-Sponsors-DS-Details.aspx

REFERENCES:
- [Derived] Barber PR, Mustapha R, Flores-Borja F, Alfano G, Ng K, Weitsman G, Dolcetti L, Suwaidan AA, Wong F, Vicencio JM, Galazi M, Opzoomer JW, Arnold JN, Thavaraj S, Kordasti S, Doyle J, Greenberg J, Dillon MT, Harrington KJ, Forster M, Coolen ACC, Ng T. Predicting progression-free survival after systemic therapy in advanced head and neck cancer: Bayesian regression and model development. Elife. 2022 Dec 23;11:e73288. doi: 10.7554/eLife.73288. PMID 36562609
- [Derived] Forster MD, Dillon MT, Kocsis J, Remenar E, Pajkos G, Rolland F, Greenberg J, Harrington KJ. Patritumab or placebo, with cetuximab plus platinum therapy in recurrent or metastatic squamous cell carcinoma of the head and neck: A randomised phase II study. Eur J Cancer. 2019 Dec;123:36-47. doi: 10.1016/j.ejca.2019.08.017. Epub 2019 Oct 21. PMID 31648099

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of 125 screened, 87 patients from 8 countries were randomized into treatment groups
Period: Overall Study
Arm/Group | Patritumab | Placebo
Started | 44 | 43
Completed | 0 | 0
Not Completed | 44 | 43
Not completed — Death | 3 | 3
Not completed — Reason not provided | 1 | 0
Not completed — Radiologic(al) progression | 23 | 23
Not completed — Clinical progression | 3 | 6
Not completed — Study terminated by sponsor | 6 | 5
Not completed — Adverse event, non-fatal | 7 | 2
Not completed — Withdrawal by Subject | 0 | 3
Not completed — Patient Request | 1 | 1

BASELINE CHARACTERISTICS:
Population: Full Analysis Set
Groups:
- Total: Total of all reporting groups
Arm/Group | Patritumab | Placebo | Total
Number analyzed (Participants) | 44 | 43 | 87
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.3 (9.18) | 61.0 (9.19) | 59.1 (9.33)
Age, Customized [Count of Participants; unit: Participants]
  18-64 Years | 32 | 27 | 59
  65-84 Years | 12 | 16 | 28
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 7 | 15
  Male | 36 | 36 | 72
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 37 | 37 | 74
  Asian | 1 | 0 | 1
  Other, Not Specified | 6 | 6 | 12
Region of Enrollment [Count of Participants; unit: Participants]
  Romania | 1 | 3 | 4
  Belgium | 1 | 1 | 2
  Hungary | 20 | 19 | 39
  Poland | 3 | 2 | 5
  United Kingdom | 9 | 5 | 14
  France | 9 | 12 | 21
  Germany | 1 | 1 | 2
Eastern Cooperative Oncology Group (ECOG) Performance Status [Count of Participants; unit: Participants]
  0=Fully active | 19 | 22 | 41
  1=Restricted in Physically Strenuous Activity | 25 | 20 | 45
  2=Ambulatory and Capable of All Self-Care | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival (PFS) in the Heregulin (HRG)-High Expression Population
Description: PFS is defined as the time from the date of randomization to the date of the first radiographic disease progression or death due to any cause, whichever comes first.
  Median PFS is from Kaplan-Meier analysis. Confidence interval (CI) for median was computed using Brookmeyer-Crowley method.
Time Frame: from Day 0 to end of active study (study termination) - within 12 months
Population: Participants in the heregulin-high expression population
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Patritumab | Placebo
Number analyzed (Participants) | 26 | 25
months | 5.56 [4.08 to 11.18] | 5.56 [3.06 to 8.29]
Statistical Analysis 1: Comparison: Patritumab vs Placebo; Heregulin-high population - Patritumab vs Placebo; Test type: Other — Both Log-rank test and Cox regression analysis did not adjust stratification factors; p = 0.8342, Log Rank — Unstratified Log-rank p-value; Hazard Ratio (HR) = 0.9291, 95% CI 2-sided [0.4856 to 1.7778]

2. Secondary Outcome: Median Overall Survival
Description: Overall survival (OS) is defined as the time from the date of randomization to death due to any cause
Time Frame: at approximately 25 months
Population: The trial terminated before sufficient data were collected for this analysis (at approximately 12 months which is prior to the time point for this analysis).
Arm/Group | Patritumab | Placebo
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Percentage of Participants With Best Overall Response
Description: Best overall response rate (ORR) is defined as the percentage of participants with Complete Response (CR) or Partial Response (PR)
Time Frame: at approximately 22 months
Population: as for outcome 2
Arm/Group | Patritumab | Placebo
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse events were collected until trial termination at 12 months.
Arm/Group | Patritumab | Placebo
All-Cause Mortality (participants affected / at risk) | 24/44 | 20/43
Serious Adverse Events (participants affected / at risk) | 19/44 | 16/43
Other Adverse Events (participants affected / at risk) | 44/44 | 42/43
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Patritumab (N=44) | Placebo (N=43)
Malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 4 (4)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Anaphylactic shock (Immune system disorders) | 0 (0) | 1 (1)
Hypersensitivity (Immune system disorders) | 1 (1) | 0 (0)
Asthenia (General disorders) | 0 (0) | 1 (1)
General physical health deterioration (General disorders) | 0 (0) | 1 (2)
Localised oedema (General disorders) | 1 (1) | 0 (0)
Non-cardiac chest pain (General disorders) | 1 (1) | 0 (0)
Malaise (General disorders) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Head Injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Ejection Fraction Decreased (Investigations) | 1 (1) | 0 (0)
Neutrophil count decreased (Investigations) | 0 (0) | 1 (1)
Weight decreased (Investigations) | 1 (1) | 0 (0)
Acute Coronary Syndrome (Cardiac disorders) | 0 (0) | 1 (1)
Arrhythmia (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac Disorder (Cardiac disorders) | 0 (0) | 1 (1)
Cardio-respiratory arrest (Cardiac disorders) | 0 (0) | 1 (1)
Cardiovascular insufficiency (Cardiac disorders) | 1 (1) | 1 (1)
Myocardial ischaemia (Cardiac disorders) | 1 (1) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Acquired tracheo-oesophageal fistula (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Lower respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0)
Loss of consciousness (Nervous system disorders) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (2)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Melaena (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Oral pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pancreatitis acute (Gastrointestinal disorders) | 0 (0) | 1 (1)
Renal failure (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal Impairment (Renal and urinary disorders) | 1 (1) | 0 (0)
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Cachexia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Decreased Appetite (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 3 (4) | 2 (2)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Arthritis bacterial (Infections and infestations) | 1 (1) | 0 (0)
Catheter site infection (Infections and infestations) | 1 (1) | 0 (0)
Device related infection (Infections and infestations) | 2 (2) | 0 (0)
Empyema (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1)
Lymphangitis (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 4 (7) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 2 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Patritumab (N=44) | Placebo (N=43)
Hypertension (Vascular disorders) | 2 (2) | 3 (4)
Hypotension (Vascular disorders) | 3 (3) | 4 (5)
Asthenia (General disorders) | 10 (14) | 11 (17)
Chills (General disorders) | 4 (5) | 2 (2)
Fatigue (General disorders) | 11 (14) | 7 (9)
Mucosal inflammation (General disorders) | 8 (13) | 2 (2)
Oedema peripheral (General disorders) | 1 (1) | 3 (3)
Pyrexia (General disorders) | 4 (7) | 1 (1)
Anxiety (Psychiatric disorders) | 2 (2) | 3 (3)
Depression (Psychiatric disorders) | 2 (2) | 3 (3)
Insomnia (Psychiatric disorders) | 4 (4) | 4 (6)
Alanine aminotransferase increased (Investigations) | 3 (6) | 2 (2)
Aspartate aminotransferase increased (Investigations) | 3 (5) | 1 (1)
Blood alkaline phosphatase increased (Investigations) | 3 (6) | 0 (0)
Neutrophil count decreased (Investigations) | 0 (0) | 3 (4)
Weight Decreased (Investigations) | 11 (16) | 10 (12)
Weight increased (Investigations) | 1 (1) | 3 (5)
Tachycardia (Cardiac disorders) | 3 (5) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 18 (34) | 13 (22)
Leukocytosis (Blood and lymphatic system disorders) | 5 (5) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 13 (23) | 11 (22)
Thrombocytopenia (Blood and lymphatic system disorders) | 10 (20) | 14 (39)
Cough (Respiratory, thoracic and mediastinal disorders) | 5 (7) | 5 (5)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 7 (12) | 5 (8)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 4 (5) | 3 (3)
Dizziness (Nervous system disorders) | 4 (4) | 2 (2)
Dysgeusia (Nervous system disorders) | 4 (4) | 0 (0)
Headache (Nervous system disorders) | 3 (4) | 5 (6)
Paraesthesia (Nervous system disorders) | 3 (3) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 4 (4) | 2 (2)
Constipation (Gastrointestinal disorders) | 7 (7) | 5 (7)
Diarrhoea (Gastrointestinal disorders) | 12 (18) | 5 (6)
Dysphagia (Gastrointestinal disorders) | 8 (10) | 4 (4)
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 4 (4) | 2 (2)
Nausea (Gastrointestinal disorders) | 16 (23) | 14 (22)
Oral Pain (Gastrointestinal disorders) | 3 (3) | 1 (1)
Stomatitis (Gastrointestinal disorders) | 5 (9) | 3 (3)
Vomiting (Gastrointestinal disorders) | 9 (11) | 7 (14)
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 15 (20) | 8 (17)
Dry skin (Skin and subcutaneous tissue disorders) | 6 (7) | 7 (8)
Pruritus (Skin and subcutaneous tissue disorders) | 3 (3) | 3 (3)
Rash (Skin and subcutaneous tissue disorders) | 20 (42) | 21 (28)
Rash Maculo-Papular (Skin and subcutaneous tissue disorders) | 3 (5) | 2 (2)
Skin fissures (Skin and subcutaneous tissue disorders) | 7 (8) | 6 (13)
Skin toxicity (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (3)
Back pain (Musculoskeletal and connective tissue disorders) | 4 (4) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 3 (6) | 4 (10)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (3)
Decreased appetite (Metabolism and nutrition disorders) | 11 (14) | 11 (17)
Hypercalcaemia (Metabolism and nutrition disorders) | 3 (3) | 3 (3)
Hypokalaemia (Metabolism and nutrition disorders) | 11 (15) | 2 (5)
Hypomagnesaemia (Metabolism and nutrition disorders) | 16 (29) | 15 (35)
Hyponatraemia (Metabolism and nutrition disorders) | 3 (4) | 1 (1)
Hypophosphataemia (Metabolism and nutrition disorders) | 2 (6) | 5 (12)
Conjunctivitis (Infections and infestations) | 6 (6) | 4 (5)
Folliculitis (Infections and infestations) | 2 (3) | 5 (6)
Paronychia (Infections and infestations) | 15 (25) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2016-06-14): https://cdn.clinicaltrials.gov/large-docs/00/NCT02633800/Prot_000.pdf
  • Statistical Analysis Plan (2016-11-29): https://cdn.clinicaltrials.gov/large-docs/00/NCT02633800/SAP_001.pdf